CLINICAL TRIAL: NCT01426958
Title: Relative Bioavailability of a Single Oral Dose of 40 mg Afatinib Given Alone Compared to Concomitant and Timed Administration of Multiple Oral Doses of Ritonavir - an Open-label, Randomised, Three-way Crossover Trial in Healthy Male Volunteers
Brief Title: Investigation of Ritonavir Effects on Afatinib Exposure in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1200.151; 2011-001803-11 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
MeSH Terms: interventions — Afatinib; Ritonavir

ARMS (3):
- treatment A (Active Comparator): 1 tablet afatinib single dose
  Interventions: Drug: afatinib
- treatment B (Experimental): 2 x 2 tablets ritonavir for 3 days + 1 tablet afatinib on the second treatment day
  Interventions: Drug: ritonavir + afatinib
- treatment C (Experimental): 2 x 2 tablets ritonavir for 3 days + 1 tablet afatinib on the second treatment day
  Interventions: Drug: ritonavir + afatinib

INTERVENTIONS:
Drug: afatinib — standard therapeutic dose
  Arms: treatment A
Drug: ritonavir + afatinib — simultaneous intake of ritonavir and afatinib on second treatment day
  Arms: treatment B
Drug: ritonavir + afatinib — on the second treatment day the first ritonavir tablet will be taken 6 hours after the afatinib tablet
  Arms: treatment C

SUMMARY:
To study the effect of the P-glycoprotein inhibitor ritonavir on the pharmacokinetics (PK) of afatinib depending on the timepoint of ritonavir administration

ELIGIBILITY:
Inclusion criteria:

1. healthy male subjects

Exclusion criteria:

1. any relevant deviation from healthy conditions

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1200.151.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: This is an open-label, randomized, three-way crossover clinical phase I trial in healthy volunteers.
Period: Overall Study
Arm/Group | All Participants
Started | 24
Completed | 22
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: This is an open-label, randomized, three-way crossover clinical phase I trial in healthy volunteers.
Arm/Group | Overall Study
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Area Under Curve From 0 to tz (AUC0-tz)
Description: AUC0-tz represents the area under the concentration curve of the analyte in plasma from 0 to the time of the last quantifiable plasma contentration of the analyte.
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96, 120 hours post
Population: This subject set includes all evaluable subjects of the treated set who were assigned to the final dose groups and who provide at least one observation for at least one primary (PK) endpoint without important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Afatinib: Subjects were treated with a single dose of Afatinib 40mg on Day 1.
- Afatinib + Concomittant Rtv: Subjects were treated with Ritonavir (Rtv) 2x100mg twice daily (bid) on Days -1, 1 and 2 and with a single dose of Afatinib 40mg on Day 1 with third Rtv dose.
- Afatinib + Timed Rtv: Subjects were treated with Rtv 2x100mg twice daily (bid) on Days -1, 1 and 2 and with a single dose of Afatinib 40mg on Day 1 six hours prior to third Rtv dose.
Arm/Group | Afatinib | Afatinib + Concomittant Rtv | Afatinib + Timed Rtv
Number analyzed (Participants) | 21 | 24 | 22
ng*h/mL | 392 (26.2) | 478 (27.9) | 438 (20.3)
Statistical Analysis 1: Comparison: Afatinib vs Afatinib + Concomittant Rtv; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.1009, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Geometric mean ratio = 119.30, 90% CI 2-sided [112.239 to 126.811], Standard Deviation 11.5 — The standard deviation is actually the geometric coefficient of variation
Statistical Analysis 2: Comparison: Afatinib vs Afatinib + Timed Rtv; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.0009, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Geometric mean ratio = 110.23, 90% CI 2-sided [103.837 to 117.006], Standard Deviation 10.9 — The standard deviation is actually the geometric coefficient of variation
Statistical Analysis 3: Comparison: Afatinib + Concomittant Rtv vs Afatinib + Timed Rtv; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.0004, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Geometric mean ratio = 91.90, 90% CI 2-sided [86.519 to 97.614], Standard Deviation 11.6 — The standard deviation is actually the geometric coefficient of variation

2. Primary Outcome: Maximum Concentration (Cmax)
Description: Cmax represents the maximum concentration of the analyte in plasma.
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96, 120 hours post
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Afatinib | Afatinib + Concomittant Rtv | Afatinib + Timed Rtv
Number analyzed (Participants) | 22 | 24 | 22
ng/mL | 19.5 (33.5) | 20.7 (29.4) | 20.7 (24.4)
Statistical Analysis 1: Comparison: Afatinib vs Afatinib + Concomittant Rtv; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.0002, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Geometric mean ratio = 104.06, 90% CI 2-sided [96.681 to 112.002], Standard Deviation 14.2 — The standard deviation is actually the geometric coefficient of variation
Statistical Analysis 2: Comparison: Afatinib vs Afatinib + Timed Rtv; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.0012, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Geometric mean ratio = 105.09, 90% CI 2-sided [96.425 to 114.530], Standard Deviation 16.1 — The standard deviation is actually the geometric coefficient of variation
Statistical Analysis 3: Comparison: Afatinib + Concomittant Rtv vs Afatinib + Timed Rtv; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.0000, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Geometric mean ratio = 99.75, 90% CI 2-sided [93.328 to 106.610], Standard Deviation 12.8 — The standard deviation is actually the geometric coefficient of variation

3. Primary Outcome: Area Under Curve From 0 to ∞ Hours (AUC0-∞)
Description: AUC0-∞ represents the area under the concentration curve of the analyte in plasma from 0 extrapolated to infinity.
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96, 120 hours post
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Afatinib | Afatinib + Concomittant Rtv | Afatinib + Timed Rtv
Number analyzed (Participants) | 22 | 24 | 22
ng*h/mL | 426 (22.8) | 515 (27.5) | 475 (19.4)
Statistical Analysis 1: Comparison: Afatinib vs Afatinib + Concomittant Rtv; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.0702, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Geometric mean ratio = 118.56, 90% CI 2-sided [111.712 to 125.822], Standard Deviation 11.5 — The standard deviation is actually the geometric coefficient of variation
Statistical Analysis 2: Comparison: Afatinib vs Afatinib + Timed Rtv; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.0005, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Geometric mean ratio = 110.76, 90% CI 2-sided [104.936 to 116.913], Standard Deviation 10.0 — The standard deviation is actually the geometric coefficient of variation
Statistical Analysis 3: Comparison: Afatinib + Concomittant Rtv vs Afatinib + Timed Rtv; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.0003, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Geometric mean ratio = 92.46, 90% CI 2-sided [86.928 to 98.341], Standard Deviation 11.9 — The standard deviation is actually the geometric coefficient of variation

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 28 days after last administration of trial medication
Arm/Group | Afatinib | Afatinib + Concomittant Rtv | Afatinib + Timed Rtv
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 2/23 | 7/24 | 5/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (N=23) | Afatinib + Concomittant Rtv (N=24) | Afatinib + Timed Rtv (N=22)
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 4
Lipase increased (Investigations) | 0 | 2 | 0
Headache (Nervous system disorders) | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.